CLINICAL TRIAL: NCT06529107
Title: Conversion of Evidence and Applied Research on Intermittent Catheterization After Radical Hysterectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West China Second University Hospital (Other)
Responsible Party: Principal Investigator, Lu Xing, deputy head nurse, West China Second University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023203
Record Dates: First submitted 2024-07-20; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Intermittent Catheterization; Conversion of Evidence

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A best evidence-based protocol for intermittent catheterization (Experimental)
  Interventions: Behavioral: intermittent catheterization protocol based on the best evidence
- Routine intermittent catheterization care (No Intervention)

INTERVENTIONS:
Behavioral: intermittent catheterization protocol based on the best evidence — A best evidence-based protocol for intermittent catheterization after radical cervical cancer surgery
  Arms: A best evidence-based protocol for intermittent catheterization

SUMMARY:
In this study, the investigators summarize the existing best evidence of intermittent catheterization in patients after radical cervical cancer surgery from the perspective of clinical translation of evidence through systematic search, evaluation and evidence integration, construct a nursing protocol of intermittent catheterization for patients after radical cervical cancer surgery based on the best evidence combined with the clinical context, and explore the clinical application effect of the above nursing protocol. It will provide a reference basis for the development of the standardization and management of intermittent catheterization for postoperative patients with cervical cancer in China, as well as the development of guidelines for intermittent catheterization after radical cervical cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≧ 18 years old
* Radical cervical cancer surgery and intermittent catheterization were performed at the Institute's hospital
* Patients or their family members can operate a smartphone
* No cognitive or psychiatric disorders, and can communicate effectively

Exclusion Criteria:

* People with serious heart, brain, lung and other important organ diseases
* People with water, electrolyte, acid-base balance disorders at the beginning of intermittent catheterization
* People with previous serious renal diseases, bladder and urethra surgery
* People with urinary tract infections
* People who did not complete all interventions or data collection
* People who voluntarily withdrew from the study or died during the study period;
* Refuse to participate in this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-10 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of urinary complications | Within 2 months of discharge
  the occurrence of urologic complications within 2 months after discharge of the patients from the hospital for follow-up, which in this study included urinary tract infections, urethral injuries, bladder stones, hydronephrosis

SECONDARY OUTCOMES:
Intermittent Catheterization Compliance Scale | Pre-intervention, immediately post-intervention, and 1 month post-discharge
  A questionnaire was used to investigate patients' adherence to carrying out intermittent catheterization before the intervention, immediately after the intervention, and 1 month after discharge from the hospital. Higher scores indicate better adherence.
12-Item Short Form Survey | Pre-intervention, immediately post-intervention, and 1 month post-discharge
  A questionnaire was used to investigate patients' quality of life before and immediately after the intervention and 1 month after discharge. Higher scores indicate better quality of life.
Self-Rating Anxiety Scale | Pre-intervention, immediately post-intervention, and 1 month post-discharge
  A questionnaire was used to investigate patients' anxiety before and immediately after the intervention and 1 month after discharge from the hospital. Higher scores indicate greater anxiety.
Intermittent Catheterization Confidence Scale | Pre-intervention, immediately post-intervention, and 1 month post-discharge
  A questionnaire was used to investigate patients' self-efficacy before and immediately after the intervention and 1 month after discharge from the hospital. Higher scores indicate greater confidence.
Utilization of health services | Within 2 months of discharge
  Follow-up to record the number of unplanned readmissions, outpatient visits, and emergency room visits within 2 months of discharge and to evaluate the patient's health service utilization

CONTACTS AND LOCATIONS:
Locations (1):
- West China Second University Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No